CLINICAL TRIAL: NCT04022928
Title: Efficacy and Safety of a Single Intraarticular Injection of Platelet-Rich Plasma on Pain and Physical Function in Patients With Ankle Osteoarthritis-a Prospective Study
Brief Title: A Single Intraarticular Injection of Platelet-Rich Plasma on Pain and Physical Function in Patients With Ankle OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Shu-Fen Sun, Director of Neutorehabilitation, MD,Department of Physical Medicine and Rehabilitation, Kaohsiung Veterans General Hospital, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS18-CT7-21
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Ankle Osteoarthritis
Keywords: Ankle joint; Osteoarthritis; Platelet rich plasma
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: patients with symptomatic ankle OA for at least 6 months were recruited. Patients received a single injection of 3-ml of PRP into symptomatic ankles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP injection (Experimental): Patients with symptomatic ankle OA for at least 6 months were recruited. Patients received a single injection of 3-ml of PRP into symptomatic ankles.
  Interventions: Other: PRP

INTERVENTIONS:
Other: PRP — , For PRP preparation, specialized platelet concentrate separator containing acid citrate dextrose as anticoagulant and a specific separator gel that harvest PR, preventing contamination of red blood cells and leukocytes were used.

SUMMARY:
Platelet-rich plasma (PRP) has been reported to be an effective treatment for knee osteoarthritis (OA). The application in ankle OA has rarely been investigated. The aim was to evaluate the efficacy and safety of a single intraarticular injection of PRP for the treatment of patients with ankle OA.

DETAILED DESCRIPTION:
Methods: In a prospective study, patients with symptomatic ankle OA for at least 6 months were recruited. Patients received a single injection of 3-ml of PRP into symptomatic ankles. The primary outcome was the change from baseline in the visual analog scale (VAS) pain score (0-10cm) at 6 months. Secondary outcomes included the Ankle Osteoarthritis Scale (AOS) score, American Orthopedic Foot and Ankle Society (AOFAS) ankle/hindfoot score, single leg stance test (SLS), use of rescue analgesics and patient satisfaction. Adverse events were recorded during the study.

Patients were followed at 1, 3 and 6 months postinjection .

ELIGIBILITY:
Inclusion Criteria:

* Age of at least twenty years
* Ankle pain lasted for at least 6 months, despite conservative treatment or inability to tolerate the side effects of medications
* Ankle radiographs taken within 6 months (reviewed by the senior author) were equivalent to grade 1-4 osteoarthritis by the Kellgren Lawrence grading system
* Average ankle pain of > 3cm on a 10-cm visual analog scale (VAS)
* Radiological evidence of bilateral ankle osteoarthritis was accepted if VAS pain in the contralateral ankle was < 3 cm
* Normal activity level, not bedridden or confined to a wheelchair, able to walk 30 meters without the aid of a walker, crutches or cane
* No use of physical therapy or changes in shoes or orthotic devices during the study

Exclusion Criteria:

* Pregnancy or lactation in women
* Lower leg trauma in a location other than within the ankle
* Previous surgery involving the spine, hip or knee
* The presence of an active infection of the ankle
* Surgery involving the affected ankle within the previous 12 months
* Intraarticular steroid or hyaluronate injection in the ankle within the previous 6 months
* Treatment with anticoagulants or immunosuppressives
* History of rheumatoid arthritis, gout, or other inflammatory arthropathy
* The presence of visual or vestibular impairments
* Poor health status (such as a neoplasm, diabetes mellitus, or paresis) that would interfere with the assessments

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) of ankle pain | 6 months
  The patient rated the average severity of ankle pain on ankle movement over the previous week on a 10-cm VAS (0=no pain to 10=worst possible pain)

SECONDARY OUTCOMES:
The Ankle Osteoarthritis Scale (AOS) score | 6 months
  AOS score is a validated patient-rated outcome measure that contains a nine-item pain subscale and a nine-item disability subscale. Using the AOS, a score of 0 represent no pain or disability and 10 represent worst pain or disability imaginable
The American Orthopedic Foot and Ankle Society (AOFAS) ankle/hindfoot score | 6 months
  a 100-point scale that devotes 40 points to pain, 50 points to function and 10 points to alignment. The maximum score of 100 points denotes no pain and normal function and alignment
The single-leg stance (SLS) test | 6 months
  SLS test involved raising the unaffected foot, without touching it to the affected lower extremity, and maintaining balance for as long as possible. Each participant performed three trials, and the best result was recorded
use of analgesic medication | through study completion, an average of 6 months
  The patient recorded the use of analgesic medication during the study period on a diary card.
global satisfaction | 6 months
  The patients rated his or her level of global satisfaction relative to the state before the treatment, using a 100 mm VAS (0= completely dissatisfied, 100=completely satisfied)
safety of PRP for ankle | through study completion, an average of 6 months
  The safety of the injection was monitored by recording the occurrence of systemic and local adverse events on a diary card

CONTACTS AND LOCATIONS:
Overall Officials: Shu Fen Sun, MD, Study Director — Kaohsiung Veterans General Hospital, Taiwan
Locations (1):
- Department of Physical Medicine and Rehabilitation, Veterans General Hospital Kaohsiung, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No